CLINICAL TRIAL: NCT05705843
Title: Intraosseous Vancomycin vs Intravenous Vancomycin in Tourniquetless Primary Total Knee Arthroplasty
Brief Title: IO vs IV Vancomycin in Tourniquetless TKA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Timothy S. Brown, Principal Investigator, The Methodist Hospital Research Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PRO00035759
Record Dates: First submitted 2023-01-19; First posted 2023-01-31 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Infection, Surgical Site
Keywords: Vancomycin; Total Knee Arthroplasty; Tourniquetless
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Intervention Model Description: This study is a prospective, randomized, single-blinded, controlled trial. The anticipated total number of participants in this study is 20 patients in each treatment arm: 20 patients will be given IV Vancomycin, 20 patients will be given IO vancomycin. This sample size is based on previous studies examining vancomycin concentration in primary TKA between IO vs IV
Who Masked: Participant, Outcomes Assessor
Masking Description: * Participant will be blinded to their mode of vancomycin administration.
  * Lab will be blinded to which group subject samples come from when doing concentration level testing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intravenous Vancomycin Administration (Active Comparator): Patients will receive the Houston Methodist Hospital orthopedic surgery standard of care pre-operative antibiotic regimen for primary total knee arthroplasty patients. This includes IV antibiotics (typically ancef or cefepime and vancomycin) will be started in the pre-operative period approximately 1 hour prior to incision (vancomycin dose weight-based at approximately 15mg/kg [12,13] generally 1000-1750mg in 500mL NS).
  Interventions: Drug: Intravenous Vancomycin
- Intraosseous Vancomycin Administration (Experimental): * IV antibiotics (per physician's standard of care): Typically ancef or cefepime is started in pre-op within 1 hour of incision. IV Vancomycin will not be administered preoperatively in this group.
  * IO vancomycin is administered via an intraosseous cannulation device (Arrow EZ-IO; Teleflex, Morrisville, NC) in the OR after sterile prep and draping has occurred prior to skin incision (500mg in 150mL NS).
  * Injection will take place into the tibial tubercle (within a pre-specified region) immediately prior to incision.
  Interventions: Drug: Intraosseous Vancomycin Injection

INTERVENTIONS:
Drug: Intraosseous Vancomycin Injection — • IO vancomycin is administered via an intraosseous cannulation device (Arrow EZ-IO; Teleflex, Morrisville, NC) in the OR after sterile prep and draping has occurred prior to skin incision (500mg in 150mL NS).
  Arms: Intraosseous Vancomycin Administration
Drug: Intravenous Vancomycin — IV Vancomycin will be started in the pre-operative period approximately 1 hour prior to incision (vancomycin dose weight-based at approximately 15mg/kg generally 1000-1750mg in 500mL NS).
  Arms: Intravenous Vancomycin Administration

SUMMARY:
Purpose of this study is to compare the efficacy of intravenous and intraosseous antibiotic administration techniques during tourniquetless total knee arthroplasty.

DETAILED DESCRIPTION:
Primary Objective: Comparable levels of vancomycin will be found in distal femur, proximal tibia, and periarticular soft tissues, as well as in systemic levels, between the intravenous and intraosseous administration groups.

Secondary Objective: Compare 30- and 90-day post-operative complication rates (infection) between the control (standard IV administration of vancomycin) versus the interventional group (intraosseous administration of vancomycin). The research team hypothesizes that there will be no difference in complication (infection) rates between groups

ELIGIBILITY:
Inclusion Criteria:

* Patient is undergoing a primary total knee arthroplasty.
* Patient is able to understand the study design and intervention and gives informed consent to participate in the study. No LAR consents will be utilized for this study.
* Age >18 years.
* Total knee arthroplasty performed without the use of a tourniquet.

Exclusion Criteria:

* Previous surgery on the knee (including arthroscopic knee surgery)
* BMI above 35
* Contraindication to receiving vancomycin, cefepime, ancef, or other standard of care pre-operative antibiotic (allergy, medical issue, etc).
* Inability to locate the tibial tubercle or administer the IO infusion
* Refusal to participate
* Uncontrolled Diabetes Mellitus type 1 or 2, defined as Hemoglobin A1C >7.5.
* Immunocompromised or immunosuppressed patients (HIV, Hep C, End-Stage Renal Disease, dialysis, transplant, chemo/radiation treatment in last 6 months, and immunosuppresive medications)

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-01-25 (Estimated); Primary Completion 2024-01-25 (Estimated); Study Completion 2024-01-25 (Estimated)

PRIMARY OUTCOMES:
Vancomycin Bone/Tissue Concentrations | immediate post-op
  Compare levels of vancomycin will be found in distal femur, proximal tibia, and periarticular soft tissues,
Systemic Vancomycin Concentrations | will be recorded day of surgery
  Compare systemic vancomycin levels between the intravenous and intraosseous vancomycin administration groups.

SECONDARY OUTCOMES:
30 day & 90 day post-operative complication rates | 30 days post-op, 90 days post-op
  Monitor charts and clinic visits during the study subject's standard of care postoperative visit schedule and monitor for adverse events including periprosthetic joint infection and wound issues.

CONTACTS AND LOCATIONS:
Locations (1):
- Houston Methodist Hospital Outpatient Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No